CLINICAL TRIAL: NCT03400813
Title: Prevention of PostConcussion-Like Symptoms for Patients Presenting at the Emergency Room: A Randomized Controlled Study of Early Single Eye Movement Desensitization and Reprocessing (EMDR) Intervention Versus Usual Care
Brief Title: Eye-Movement Desensitization and Post-Traumatic Syndroms
Acronym: SOFTER3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Centre Hospitalier de Cadillac (Other); Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHUBX 2017/13
Record Dates: First submitted 2017-11-20; First posted 2018-01-17 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Post-Concussion Symptoms; Post-Traumatic Stress Disorder
Keywords: Eye-Movement Desensitization; Reprocessing
MeSH Terms: conditions — Post-Concussion Syndrome; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator / Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients in this group continue their usual care without intervention.
- R-TEP EMDR (Experimental): Patients in R-TEP EMDR group will receive the intervention.
  Interventions: Behavioral: R-TEP EMDR

INTERVENTIONS:
Behavioral: R-TEP EMDR — Recent Traumatic Episode Protocol Eye-Movement Desensitization and Reprocessing is a early and short adaption protocol of EMDR developed by Shapiro E. EMDR is a psychotherapeutic approach that can rapidly process disturbing experiences adaptively together with the aid of eye movements or other forms of bi-lateral stimulation.
  Arms: R-TEP EMDR

SUMMARY:
Millions people, all over the world, are admitted in the Emergency Department after a trauma or simply to receive medical cares. In France, it represents 10 million patients. Probably because of stress associated with the event, 20% will suffer a combination of non-specifics symptoms which persist for many months and with daily life quality impairment. The investigators hypothesize that an early intervention, such as Eye-Movement, Desensitization and Reprocessing (EMDR) could be performed in the ED and could prevent the occurrence of these symptoms.

DETAILED DESCRIPTION:
Emergency department are a privileged service for patients suffering from trauma and stressful medical conditions. In France, every year 10 million people come or are taken to the emergency department (ED). Many studies have shown that 10-20% of these trauma patients develop a non-specific set of symptoms that can persist for several months after ED assessment. These includes, for example, headache, memory and/or concentration impairment, stress intolerance, irritability... These symptoms lead to an alteration in the quality of social, family and professional life, and therefore affect one to two millions people in France alone.

The association between these symptoms and mild traumatic brain injury (MTBI) has already been demonstrated. It was defined as post-concussion syndrome (PCS) according to the DSM-IV-TR. However, several recent studies have shown that these symptoms are not specific to MTBI but may appear for any type of trauma and event for stressful medical conditions. PCS seems to appear for events occurring in a stressful environment or in people with psychological weaknesses. These symptoms will therefore be referred here to Post-concussion-like symptoms (PCLS). Moreover, PCLS appear to be very similar and sometime overlap those of the numbing and hyperarousal dimension of the Post Traumatic Stress Disorder (PTSD).

A recent study, carried out by our team in the ED of Bordeaux University Hospital, showed that PCLS was associated with a high level of stress at ED discharge, whatever that stress level at entry.

The Eye-Movement Desensitization and Reprocessing (EMDR) is a recognized psychotherapeutic approach in the treatment of PTSD and several single-session versions of the protocol have been proposed : one of them is Recent Traumatic Episode Protocol EMDR (R-TEP EMDR).The investigators hypothesize that the introduction of an early R-TEP EMDR intervention in emergencies can reduce the level of stress and thus the occurrence of the PCLS and PTSD symptoms among a subset of patients screened for their high risk of PCLS.

The study is a two-site open-label two-group randomized controlled trial designed to assess the efficacy of an early R-TEP EMDR intervention performed in the ED by comparing PCLS and PTSD symptoms at 3 and 12 months between the two randomization groups: (i) R-TEP EMDR; (ii) care as usual.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in department (i) injured whatever the cause of injury. The event causing the injury must have occurred in the past 12 hours; or (ii) experiencing a medical event associated with a medical acute condition and presenting for the first time at the ED for this motive
* Score resulting from the screening tool>= 2 : Female gender: +1 Taking at least one anxiolytic treatment: + 1 Perceived health status prior to admission: Excellent, very good: 0 ; Good: +1 Poor: +2 ; Bad: +3
* Affiliated to French insurance system.

Exclusion Criteria:

* Refusal to participate in the study
* Current drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Inability to answer questionnaire: any cognitive impairement, language barrier, consciousness disorder...
* Impossibility of recontacting the patient at a distance from the trauma (no telephone contact ...)
* Patient already included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Compare the impact on 3-months PostConcussion-Like Syndrome (PCLS) of early Early EMDR R-TEP | 3 months after inclusion visit
  3-months PCLS as measured with the Rivermead Postconcussion Symptoms Questionnaire

SECONDARY OUTCOMES:
Recovery expectation at discharge following participant' recruitment | 3 months after inclusion visit
  Self-reported to ER medical staff thanks to a Rivermead questionnaire
Acute pain | 3 months after inclusion visit
  Self-reported acute pain to ER medical staff using the total score of a 10 points Likert scale
Chronic pain | 3 months after inclusion visit
  chronic pain will be self-reported thanks to a Rivermead questionnaire
Psychotropic medicines use | 3 months after inclusion visit
  Psychotropic medicines use will be measured by drug delivery data as extracted from the Caisse national d'assurance maladie des travailleurs salariés (CNAM-TS) database, the French social insurance system.
Compare the impact on 12-months PostConcussion-Like Syndrome (PCLS) of early Early EMDR R-TEP. | 12 months after inclusion visit
  12-months PCLS as measured with the the Rivermead Postconcussion Symptoms Questionnaire
Compare the impact on 3-months Post-Traumatic Stress Disorder (PTSD) of early EMDR R-TEP. | 3 months after inclusion visit
  3-months PTSD as measured with PTSD Checklist-5

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Lagarde, PhD, Study Director — University Hospital Bordeaux, France
Locations (2):
- France (2):
  - Emergency department, Bordeaux University Hospital, Bordeaux
  - University Hospital, Lyon, Lyon

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Gil-Jardine C, Al Joboory S, Jammes JTS, Durand G, Ribereau-Gayon R, Galinski M, Salmi LR, Revel P, Regis CA, Valdenaire G, Poulet E, Tazarourte K, Lagarde E. Prevention of post-concussion-like symptoms in patients presenting at the emergency room, early single eye movement desensitization, and reprocessing intervention versus usual care: study protocol for a two-center randomized controlled trial. Trials. 2018 Oct 12;19(1):555. doi: 10.1186/s13063-018-2902-2. PMID 30314512